CLINICAL TRIAL: NCT06168344
Title: The Effect of Web-Based Education Given to Mothers of Infants With Congenital Heart Disease on Quality of Life and Self Efficacy
Brief Title: The Effect of Web-based Training Given to Mothers of Babies With Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Berna Eren Fidancı, Associate professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GHF_NU1
Record Dates: First submitted 2023-11-02; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Mothers; Quality of Life; Self Efficacy; Training
Keywords: Congenital Heart Disease; Web-Based Education; Mothers; Infants; Care; Pediatric Nursing
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: There are two groups in the study. Web-based education was provided to mothers in the intervention group (n=30). No intervention was applied to the mothers in the control group (n=30) other than the outpatient clinic routine of the hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Mothers were assigned to groups by simple randomization method. The website was designed, mothers were given their usernames and passwords and their memberships were created. Pretests (Parent-Baby Introductory Information Form, Quality of Life Scale and Generalized Perceived Self-Efficacy Scale) were administered via the website. Mothers completed the modules in the web-based training program within four weeks. Four weeks later, posttests (Quality of Life Scale and Generalized Perceived Self-Efficacy Scale) were administered via the website.
  Interventions: Other: Web-Based Education Program
- Control Group (No Intervention): Mothers' usernames and passwords were created and website memberships were made. Pretests (Parent-Baby Introductory Information Form, Quality of Life Scale and Generalized Perceived Self-Efficacy Scale) were applied. Website use by mothers in the control group was restricted and access to web-based educational content was closed to all mothers in this group. The mothers in the control group were applied the hospital outpatient clinic routine without any intervention. Four weeks later, posttests (Quality of Life Scale and Generalized Perceived Self-Efficacy Scale) were administered via the website. Pre-test and post-tests of mothers in the control group were collected via the website. After the research data was collected, a web-based training program was opened to the mothers in the control group and they were allowed to benefit from the training content.

INTERVENTIONS:
Other: Web-Based Education Program — This study was assessed the impact of a web-based education program provided to mothers of infants with congenital heart diseases on their quality of life and self-efficacy levels
  Arms: Intervention Group

SUMMARY:
This study was assessed the impact of a web-based education program provided to mothers of infants with congenital heart diseases on their quality of life and self-efficacy levels. The study is a mixed-method approach with a qualitative and pre-test post-test design, utilizing randomized controlled quasiexperimental type.

The research was conducted with mothers of infants diagnosed with congenital heart disease who sought care at the Pediatric Cardiology Outpatient Clinic of a university hospital and were followed up. There are two groups in the study. Web-based education was provided to mothers in the intervention group (n=30). No intervention was applied to the mothers in the control group (n=30) other than the outpatient clinic routine of the hospital.

DETAILED DESCRIPTION:
Materials and Methods: study is a mixed-method approach with a qualitative and pre-test post-test design, utilizing randomized controlled quasiexperimental type. The research was conducted with mothers of infants diagnosed with congenital heart disease who sought care at the Pediatric Cardiology Outpatient Clinic of a university hospital and were followed up. There are two groups in the study. Web-based education was provided to mothers in the intervention group (n=30). No intervention was applied to the mothers in the control group (n=30) other than the outpatient clinic routine of the hospital. "Qualitative interview form, Parent-infant Introductory Information Form, Quality of Life Scale and Generalized Perceived Self-Efficacy Scale" were used. The research process had two stages; in the first stage, qualitative data was collected and after qualitative interviews with mothers, the content of the web-based training was created in line with the needs of the mothers. In the second stage, quantitative data were collected, and a web-based training program was applied to the intervention group and an outpatient clinic routine to the control group.

ELIGIBILITY:
Inclusion Criteria:

* For mothers;
* Having a baby with congenital heart disease
* Being over 18 years of age
* Being literate
* Being able to speak and understand Turkish
* There is no health problem that may prevent participation in training.
* Being able to use a computer/mobile phone
* Being able to use and have internet access
* Volunteering to participate in research

For babies;

* Those born at or after the 37th week of gestation and those with congenital heart disease, aged 0-12 months
* Has not had heart surgery
* Babies who do not have any other chronic diseases

Exclusion Criteria:

* Filling out forms incompletely
* Being a foreign national
* Having vision or hearing problems
* To give up participating in the research
* Mothers and babies who have physical/mental problems that may affect the research results during the study period.

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Qualitative Interview Form | In the first stage of the research; Qualitative data were collected: once
  In the first stage of the research; Qualitative data were collected. Qualitative interviews were conducted with mothers (n=11). Seven open-ended questions were asked. Categories and themes were arranged according to the content analysis created from the data. The content of the Web-based training program was created in line with the needs and requirements of mothers according to categories and themes.

SECONDARY OUTCOMES:
Parent-Baby Identification Information Form | Form was administered to mothers in both groups before the study: once.
  The form consists of a total of 23 questions and two sections. The first part consists of 14 questions to evaluate the socio-demographic characteristics of parents. Second part consists of nine questions to evaluate the demographic characteristics of babies.

OTHER OUTCOMES:
Quality of Life Scale Short Form (SF-36) | SF-36 was applied to mothers in the intervention and control groups: pretest-posttest, twice (15 minutes)
  SF-36 is a 36-question measurement tool that examines eight dimensions of health-related quality of life.
Generalized Perceived Self-Efficacy Scale (GASS) | GASS was applied to mothers in the intervention and control groups: pretest-posttest, twice (15 minutes)
  GASS is a 10-item scale that measures the self-efficacy level of mothers

CONTACTS AND LOCATIONS:
Overall Officials: Berna EREN FİDANCI, Assoc. Prof., Study Director — University of Saglik Bilimleri
Locations (1):
- Eskişehir Osmangazi University Health Practice and Research Hospital, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes